CLINICAL TRIAL: NCT02710799
Title: Evaluation of the Effectivity of Teleconsultations for Improving the Referrals From Primary Care to Specialized Care of Patients With Chronic Endocrinological Conditions
Brief Title: Evaluation of the Effects of Teleconsultations on a Endocrinology Referral List
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Secretaria Estadual da Saúde do Estado do Rio Grande do Sul (Unknown); Programa de Pesquisa e Pós-Graduação em Epidemiologia da UFRGS (Unknown); TelessaúdeRS / UFRGS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 32981014.0.0000.5327; U1111-1179-2949 (Registry Identifier: UTN)
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus; Hypothyroidism; Hyperthyroidism; Goiter; Thyroid Nodule; Obesity
Keywords: Endocrinology; Referral list; Teleconsultation; Telemedicine; Cluster randomized clinical trial
MeSH Terms: conditions — Diabetes Mellitus; Hypothyroidism; Hyperthyroidism; Goiter; Thyroid Nodule; Obesity | interventions — Remote Consultation; Clinical Protocols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Referrals will be evaluated through the state's protocols
  Interventions: Other: Protocol
- Intervention (Experimental): Referrals will be evaluated through the state's protocols associated with telephone-based teleconsultations.
  Interventions: Other: Teleconsultation; Other: Protocol

INTERVENTIONS:
Other: Teleconsultation — The teleconsultations will be performed by medical doctors, mostly family physicians, but also internists and endocrinologists. The teleconsultations will follow a structured format to discuss some topics on the disease and access the relevant information (based on the state's protocols). The doubts from the primary care physician will be addressed.
  Arms: Intervention
Other: Protocol — The informations provided in the referral list will be evaluated through the state's referrals protocols.

SUMMARY:
The aim of this study is evaluate the effects of telephone teleconsultations to primary care physicians (compared to the state's referral protocol) in the referrals waiting list for endocrinological appointments.

DETAILED DESCRIPTION:
Rio Grande do Sul state's referral list for endocrinology evaluation in specialized care is highly overloaded. There is currently a referral protocol to select patients how should be referred. It will be evaluated if a intervention of telephone-based teleconsultations provided by the TelessaúdeRS to the primary care physicians can provide additional benefits. TelessaúdeRS is a telehealth program from the University of Rio Grande do Sul. This will be evaluated in a cluster randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients from counties with at least 5 endocrinology referrals waiting appointment.
* Patients referred from primary care physicians
* Patients referred because one of the protocol conditions (Diabetes Mellitus, Hypothyroidism, Hyperthyroidism, Goiter, Thyroid nodule, Obesity).

Exclusion Criteria:

* Patients from counties with more than one hundred endocrinology referrals waiting appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3470 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of consultations authorized | 1 year
  Number of consultations authorized after the evaluation by the control and intervention strategies.

SECONDARY OUTCOMES:
Number of new referrals for endocrinology | 1 year
  Total number of new referrals performed by the county.
Adherence to the state's protocols | 1 year
  Number of new referrals for endocrinology with adequate informations according to the state's protocols.
Usage of TelessaúdeRS teleconsultations | 1 year
  Total number of calls to TelessaúdeRS hotline (available to every primary care physician working in brazilian public health system)

CONTACTS AND LOCATIONS:
Overall Officials: Erno Harzheim, MD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Secretaria Estadual da Saúde, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We plan to publish trial results in an indexed medical journal. The results will be reported by the authors and the authorship criteria from ICMJE will be followed. After publishing the main results of the trial the unidentified dataset will be available by contacting the authors and providing an analyses plan which will be evaluated by the study's main investigator.